CLINICAL TRIAL: NCT05396170
Title: Phlebotomy in Blood Donors and Polycythemia Vera Patients- The Effect on Physiology: An Orienting Case-Cross Over Study
Brief Title: Effect of Phlebotomy on Heartrate in Polycythemia Patients
Acronym: NOSFERATU
Status: Recruiting | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, jjzwaginga, Prof. dr. J.J. Zwaginga, Leiden University Medical Center
Other Study IDs: N22.055
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Polycythemia
MeSH Terms: conditions — Polycythemia | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: phlebotomy — 500ml of blood phlebotomized per standard of care to reduce symptoms from polycythemia

SUMMARY:
Single-centre, observational within-subject design: patients that undergo phlebotomies regularly for polycythemia will be measured continuously by wearables one week before until one week after a phlebotomy, for three phlebotomies.

DETAILED DESCRIPTION:
Rationale: Little is known about the effect of a hemoglobin-shift on patients, anaemic, non-anaemic or even polycythaemic. It has been established that severe anaemia has deteriorating effects on the patient, which can be (partially) reversed by treatments like transfusion, erythropoietin stimulating agents or iron/vitamin supplements, depending of the etiology of the anaemia. However, the optimal haemoglobin target and threshold for such treatments has yet to be determined. It is therefore necessary to evaluate what the exact effect of various haemoglobin levels, and a shift therein, is on the physiology of patients. Only then can the benefits be weighed properly against the risks for individual patients when considering treatment for anaemia, safety of blood donation, or expected effect of phlebotomy for polycythaemia.

Primary Objective:

- Compare the per individual and per group effects of a reduction in Hb mass on physical functional outcomes (heart rate; activity parameters; QoL) in patients with polycythaemia.

Secondary Objectives:

- Compare the primary outcomes to data from the REMOTE-2 and FAINT-study (similar measurements in transfusion dependent patients and whole blood donors)

Study design: Within-subject design. Patients will be remotely monitored one week before phlebotomy until one week after.

Study population: Adult patients with a polycythaemia requiring phlebotomies on a regular basis.

Main study parameters: heart rate, blood pressure, activity parameters and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with polycythaemia, requiring phlebotomy on a regular basis (at least every 4 months)
* Subjects aged ≥18 years
* In possession of a smartphone
* Life expectancy ≥ 3 months

Exclusion Criteria:

* Poor performance/functional status (Eastern Cooperative Oncology Group system ECOG ≥3)
* Participants with known arrhythmias or other significant cardiological conductivity disorders (Paroxysmal atrial fibrillation is allowed)
* Hospitalized subjects
* Subjects with a pacemaker.
* Subjects with a secondary polyglobulia due to eg smoking or other pulmonary issues.
* Scheduled oncological treatments or surgery during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with polycythaemia, requiring phlebotomy on a regular basis (at least every 4 months)
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2022-07-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Mean heart rate as measured by the withings BPM and withings Steel HR biodevices | one week before until one week after phlebotomy; for three phlebotomies
  the Withings BPM will give point measurements while the withings Steel HR gives continuous heart rate measurements. We will compare before the phlebotomy to after phlebotomy and >48hrs after phlebotomy, within-subjects.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure as measured by the withings BPM connect. | Daily basis from one week before until one week after phlebotomy; three phlebotomies
  BP (systolic/diastolic) measured by Withings BPM connect
Number of steps per 24hrs as measured by the withings steel HR | one week before until one week after phlebotomy; for three phlebotomies
  Steps as a measure for activity as measured by the withings steel HR
Quality of life as measured by the EuroQol-5D questionnaire (EQ5D) | Daily basis from one week before until one week after phlebotomy; three phlebotomies
  QoL as measured by the castor-based EQ5D. The EQ5D gives two scores: the utility score (range: -.329 to 1, higher is better, lower than 0 is considered worse than death) and an VAS (visual analogue scale) score (range 0 to 100, higher is better)

CONTACTS AND LOCATIONS:
Overall Officials: Jaap Jan Zwaginga, MD, PhD, Principal Investigator — LUMC
Locations (1):
- LUMC, Leiden, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Stored in non-publicly available repository, will be made available on request
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After completion of trial
Access Criteria: available on request by contacting coordinating researcher

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT05396170/Prot_SAP_000.pdf